CLINICAL TRIAL: NCT05702476
Title: Marfan Syndrome (MFS) and Facial Dysmorphism: Non-invasive 3D Assessment
Acronym: FACE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: FACE
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Rare Diseases; Marfan Syndrome
Keywords: Rare Diseases; Marfan syndrome; Facial features
MeSH Terms: conditions — Rare Diseases; Marfan Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MFS Adult patients: Patients with clinical and/or gentic diagnosis of MFS older than 18 years
- MFS Paediatric patients: Patients with clinical and/or gentic diagnosis of MFS younger than 18 years

SUMMARY:
The goal of this study observational prospective study is to define the facial morphological features associated with Marfan syndrome (MFS). The main qustion it aims to answer are:

1. To describe the facial morphological features associated with MFS and their evolution over time;
2. To study the association between facial morphology and the features of reference for the diagnosis of MFS.

DETAILED DESCRIPTION:
Marfan syndrome (MFS, OMIM # 154700) is a rare connective tissue disorder caused by mutations in the gene encoding fibrillin-1 glycoprotein (FBN1), involved in the development of microfibrils. Since FBN1 is a constituent of the connective tissue present at a systemic level, mutations in its gene lead to alterations of the connective tissue, even with pleiotropic effects. The clinical manifestations of MFS are heterogeneous and can occur at any time, from neonatal onset to infancy or adolescence. In this sense, the presence of facial dysmorphism could help in early diagnosis of the disease. Considering the craniofacial features, the phenotypic manifestation related to the syndrome MFS are: dolichocephaly, eyelid down-slanting, malar hypoplasia and retrognathia. However, Few studies have so far studied the facial features associated with MFS. Morevoer, there is a gap in the literature for the evaluation of the progression of facial morphology in the pediatric MFS population as well as potential correlations between facial dysmorphism and other manifestations of the disease.

ELIGIBILITY:
Inclusion Criteria:

* White european ethnicity;
* Signed informed consent;

Exclusion Criteria:

* Previous relevant traumas affecting the craniofacial district or maxillofacial surgery;
* Presence of beard and mustache;
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinical and/or genetic diagnosis of MFS currently in follow-up at Cardiovascular Genetic Cenrte, IRCCS Policlinico San Donato.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Disease Progression | 18 months
  Prospective evaluation focused in the craniofacial area in MFS patients

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pini, MD, Principal Investigator — Cardiovascular-Gentic Centre, IRCCS Policlinico San Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Lombardy, Italy